CLINICAL TRIAL: NCT05736939
Title: Gender Differences in the Recovery Rate Following a Hybrid Pulmonary Rehabilitation Programme in Patients With Long COVID-19 Syndrome
Brief Title: Gender Differences in the Recovery Rate Following PR in Patients With Long COVID-19
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Nikolaos Chynkiamis, Clinical Exercise Physiologist, National and Kapodistrian University of Athens
Other Study IDs: 24633
Record Dates: First submitted 2023-02-19; First posted 2023-02-21 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Post Acute COVID-19 Syndrome
Keywords: Post-Acute COVID-19 Syndrome; Pulmonary Rehabilitation; Muscle strength; Quality of life
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men with long COVID-19 syndrome: Patients were male adults (>18 years), with persistent symptoms more than 3 months since the acute phase of the COVID-19.
  Interventions: Other: Out-patient Pulmonary Rehabilitation
- Women with long COVID-19 syndrome: Patients were women adults (>18 years), with persistent symptoms more than 3 months since the acute phase of the COVID-19.
  Interventions: Other: Out-patient Pulmonary Rehabilitation

INTERVENTIONS:
Other: Out-patient Pulmonary Rehabilitation — Pulmonary Rehabilitation (PR) programme consisting of 30 minutes interval aerobic exercise on cycle ergometers at 100% of peak work rate (WRpeak) and resistance exercises for the upper body. Dyspnoea and leg discomfort were recorded on the modified 1-10 Borg scale, whereas heart rate (HR) and oxygen saturation (SpO2%) were monitored by a pulse oximeter. Based on symptoms of breathlessness and fatigue reported at the end of each session, the exercise intensity was increased by 5-10% of the baseline WRpeak in the next session. The remote 24 home-based PR sessions consisted of 30 minutes walking with an individualised target of steps, recorded via the mobile app installed in the patients' mobile phone. The steps, leg discomfort and dyspnoea were reported by the patient via a physical activity diary on a weekly basis. If dyspnoea and fatigue were both <4 at the Borg scale the weekly target of steps was increased by 5-10% by the assessors.

SUMMARY:
The goal of this retrospective analysis is to compare the magnitude of improvement in respiratory and peripheral muscle strength, following the completion of a hybrid pulmonary rehabilitation programme, in men and women with long COVID-19 syndrome. The main question it aims to answer is the following:

• does gender limits the effects of a hybrid pulmonary rehabilitation programme on respiratory and peripheral muscle strength?

DETAILED DESCRIPTION:
As of January 2023, more than 500 million people have been affected by Severe Acute Respiratory Distress Syndrome-Coronavirus-2 (SARS-COV-2) globally. In Greece, since January 2020 there have been more than 5 million confirmed cases of COVID-19 and more than 35,000 deaths. Based on this data, it seems that the majority of patients recover (even those requiring hospital admission) but present with persistent symptoms at least three months after the acute illness, a condition defined as 'Long COVID-19'. The most commonly reported symptoms include long-standing fatigue, dyspnoea, muscle and joint pain, sleep disturbances, short-term memory loss and brain fog.

This syndrome affects a large group of patients, and according to World Health Organisation it imposes a great burden on the healthcare systems worldwide. Consequently, it is important to identify preventable risk factors for 'Long COVID-19' in order to address the complex needs of these patients and reduce the prevalence of this new long-term condition.

According to the Post-hospitalisation COVID-19 study (PHOSP-COVID) which has included adults with COVID-19 discharged from United Kingdom hospitals, the main risk factors associated with worse recovery at 1 year involved obesity, need for invasive mechanical ventilation during the acute illness and female sex. Other studies evaluating the prevalence of 'Long COVID-19' in the two sexes found that female patients were more likely to have one or more symptoms 12 months following the acute phase of the disease. Despite the fact that lengths of hospital and ICU stay were reduced in women compared to men, female sex proved to be an independent risk factor for the development of ongoing symptoms, among which were fatigue, dyspnoea, muscle aches and generalised weakness. The autoimmune hypothesis could account for the higher incidence of 'Long COVID-19' syndrome in women. According to this hypothesis, the immune response for both genetic and hormonal factors is stronger in women compared to men and hence autoimmune reactions are more prevalent in women.

Guidelines have been published suggesting the implementation of pulmonary rehabilitation (PR) programmes for the management of patients with 'Long COVID-19' syndrome. According to recently published systematic reviews, pulmonary rehabilitation is beneficial for patients with long COVID-19 syndrome in terms of quality of life, muscle strength, walking capacity and sit-to-stand performance. Whether reduced recovery prognosis and long-lasting ongoing symptoms in women adversely affect the outcome of rehabilitation is still unknown. This is an important issue for healthcare systems when considering management strategies for people with 'Long COVID-19' syndrome. Furthermore, tele-rehabilitation programmes are feasible and effective in improving physical capacity, quality of life and symptoms in adult survivors of COVID-19.

Accordingly, the present study looked into the effect of a hybrid rehabilitation programme (including out-patient and home-based sessions) on physical and mental health outcomes in previously hospitalised women and men with 'Long COVID-19' syndrome. It was hypothesised that the magnitude of improvement in women would be less compared to men.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation due to Sars-COV-2 infection.
* Presence of persistence fatigue assessed via FACIT questionnaire.

Exclusion Criteria:

Exclusion criteria include presence of any of the following list within 3 months prior to informed consent:

* participation in another clinical trial
* occurrence of myocardial infarction
* hospitalisation for unstable angina
* stroke
* coronary artery bypass graft (CABG)
* percutaneous coronary intervention (PCI)
* implantation of a cardiac resynchronisation therapy device (CRTD)
* active treatment for cancer or other malignant disease
* uncontrolled congestive heart disease (NYHA class >3)
* acute psychosis or major psychiatric disorders or continued substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Τhe study population consists of patients who have been diagnosed with long COVID-19 based on the persistence of fatigue at least three months following hospital discharge due to COVID-19. All patients participated in a pulmonary rehabilitation programme which is provided in these patients by our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Fatigue | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Degree of fatigue will be assessed via the Functional Assessment of Chronic Illness Therapy questionnaire

SECONDARY OUTCOMES:
Quadriceps muscle strength | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Quadriceps muscle strength will be reported as maximum strength in kg
Handgrip muscle strength | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Handgrip muscle strength will be reported as maximum strength in kg
Inspiratory muscle strength | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Inspiratory muscle strength will be reported as maximum strength in centimeters water
Expiratory muscle strength | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Expiratory muscle strength will be reported as maximum strength in centimeters water
Dyspnoea | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Dyspnoea will be assessed via completion of modified Medical Research Council Dyspnoea Scale questionnaire. The score ranges from 0-4. The greater the score, the worse the dyspnoea levels
Emotional status | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Emotional status will be assessed via completion of the Hospital Anxiety and Depression. Scale questionnaire. The score ranges from 0-21 for each component (anxiety and depression). The higher the score, the higher the levels of anxiety and depression.
Symptoms | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Symptoms will be assessed via completion of the Chronic Obstructive Pulmonary Disease Assessment Tool questionnaire. The score ranges from 0-40 points. The higher the score, the worse the prognosis.
Self-reported quality of life | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Self-reported quality of life will be assessed via completion of the EuroQol-5Dimension-5Levels questionnaire.
Post traumatic stress disorder (PTSD) | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  PTSD will be assessed via completion of the Impact Event Scale-Revised questionnaire.The total score ranges from 0-88. The higher the score, the higher the levels of PTSD
Six minute walk distance covered | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  The distance that patients cover during the six minute walk test.
Short Physical Performance Buttery test (SPPB) | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  SPPB is a series of test including balance, 4 meter walk and 5 sit-to-stand repetitions. The test assess the functional capacity of the patients.
Level of daily physical activity | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Level of daily physical activity will be reported as steps per day the week prior the initiation of the intervention and one week following the completion of the intervention.
Exercise tolerance | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Exercise tolerance will be assessed by performing a cardiopulmonary exercise test.
Cardiac function | Prior and following the completion of a 3 month pulmonary rehabilitation programme (At 0 and at 3 months)
  Cardiac function will be assessed via a resting echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Chynkiamis, Ph.D., Principal Investigator — Sotiria General Hospital for Chest Diseases, Athens, Greece
Locations (1):
- Sotiria Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared to any other research team. The data that will be collected retrospectively for the present study as the patients have already completed the pulmonary rehabilitation programme. The rehabilitation department of our clinic is responsible for the storage and the management of patients data. In that content, they will share with the research team the necessary data to complete our study. The research team is not authorised to share the data with other research teams or researchers.

REFERENCES:
- [Background] Goertz YMJ, Van Herck M, Delbressine JM, Vaes AW, Meys R, Machado FVC, Houben-Wilke S, Burtin C, Posthuma R, Franssen FME, van Loon N, Hajian B, Spies Y, Vijlbrief H, van 't Hul AJ, Janssen DJA, Spruit MA. Persistent symptoms 3 months after a SARS-CoV-2 infection: the post-COVID-19 syndrome? ERJ Open Res. 2020 Oct 26;6(4):00542-2020. doi: 10.1183/23120541.00542-2020. eCollection 2020 Oct. PMID 33257910
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Evans RA, McAuley H, Harrison EM, Shikotra A, Singapuri A, Sereno M, Elneima O, Docherty AB, Lone NI, Leavy OC, Daines L, Baillie JK, Brown JS, Chalder T, De Soyza A, Diar Bakerly N, Easom N, Geddes JR, Greening NJ, Hart N, Heaney LG, Heller S, Howard L, Hurst JR, Jacob J, Jenkins RG, Jolley C, Kerr S, Kon OM, Lewis K, Lord JM, McCann GP, Neubauer S, Openshaw PJM, Parekh D, Pfeffer P, Rahman NM, Raman B, Richardson M, Rowland M, Semple MG, Shah AM, Singh SJ, Sheikh A, Thomas D, Toshner M, Chalmers JD, Ho LP, Horsley A, Marks M, Poinasamy K, Wain LV, Brightling CE; PHOSP-COVID Collaborative Group. Physical, cognitive, and mental health impacts of COVID-19 after hospitalisation (PHOSP-COVID): a UK multicentre, prospective cohort study. Lancet Respir Med. 2021 Nov;9(11):1275-1287. doi: 10.1016/S2213-2600(21)00383-0. Epub 2021 Oct 7. PMID 34627560
- [Background] PHOSP-COVID Collaborative Group. Clinical characteristics with inflammation profiling of long COVID and association with 1-year recovery following hospitalisation in the UK: a prospective observational study. Lancet Respir Med. 2022 Aug;10(8):761-775. doi: 10.1016/S2213-2600(22)00127-8. Epub 2022 Apr 23. PMID 35472304
- [Background] Wynberg E, van Willigen HDG, Dijkstra M, Boyd A, Kootstra NA, van den Aardweg JG, van Gils MJ, Matser A, de Wit MR, Leenstra T, de Bree G, de Jong MD, Prins M; RECoVERED Study Group. Evolution of Coronavirus Disease 2019 (COVID-19) Symptoms During the First 12 Months After Illness Onset. Clin Infect Dis. 2022 Aug 24;75(1):e482-e490. doi: 10.1093/cid/ciab759. PMID 34473245
- [Background] Thompson EJ, Williams DM, Walker AJ, Mitchell RE, Niedzwiedz CL, Yang TC, Huggins CF, Kwong ASF, Silverwood RJ, Di Gessa G, Bowyer RCE, Northstone K, Hou B, Green MJ, Dodgeon B, Doores KJ, Duncan EL, Williams FMK; OpenSAFELY Collaborative; Steptoe A, Porteous DJ, McEachan RRC, Tomlinson L, Goldacre B, Patalay P, Ploubidis GB, Katikireddi SV, Tilling K, Rentsch CT, Timpson NJ, Chaturvedi N, Steves CJ. Long COVID burden and risk factors in 10 UK longitudinal studies and electronic health records. Nat Commun. 2022 Jun 28;13(1):3528. doi: 10.1038/s41467-022-30836-0. PMID 35764621
- [Background] Boscolo-Rizzo P, Guida F, Polesel J, Marcuzzo AV, Capriotti V, D'Alessandro A, Zanelli E, Marzolino R, Lazzarin C, Antonucci P, Sacchet E, Tofanelli M, Borsetto D, Gardenal N, Pengo M, Tirelli G. Sequelae in adults at 12 months after mild-to-moderate coronavirus disease 2019 (COVID-19). Int Forum Allergy Rhinol. 2021 Dec;11(12):1685-1688. doi: 10.1002/alr.22832. Epub 2021 Jun 9. No abstract available. PMID 34109765
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Lindahl A, Aro M, Reijula J, Makela MJ, Ollgren J, Puolanne M, Jarvinen A, Vasankari T. Women report more symptoms and impaired quality of life: a survey of Finnish COVID-19 survivors. Infect Dis (Lond). 2022 Jan;54(1):53-62. doi: 10.1080/23744235.2021.1965210. Epub 2021 Aug 19. PMID 34410220
- [Background] Fernandez-de-Las-Penas C, Martin-Guerrero JD, Pellicer-Valero OJ, Navarro-Pardo E, Gomez-Mayordomo V, Cuadrado ML, Arias-Navalon JA, Cigaran-Mendez M, Hernandez-Barrera V, Arendt-Nielsen L. Female Sex Is a Risk Factor Associated with Long-Term Post-COVID Related-Symptoms but Not with COVID-19 Symptoms: The LONG-COVID-EXP-CM Multicenter Study. J Clin Med. 2022 Jan 14;11(2):413. doi: 10.3390/jcm11020413. PMID 35054108
- [Background] Brodin P. Immune determinants of COVID-19 disease presentation and severity. Nat Med. 2021 Jan;27(1):28-33. doi: 10.1038/s41591-020-01202-8. Epub 2021 Jan 13. PMID 33442016
- [Background] Spruit MA, Holland AE, Singh SJ, Tonia T, Wilson KC, Troosters T. COVID-19: interim guidance on rehabilitation in the hospital and post-hospital phase from a European Respiratory Society- and American Thoracic Society-coordinated international task force. Eur Respir J. 2020 Dec 3;56(6):2002197. doi: 10.1183/13993003.02197-2020. Print 2020 Dec. PMID 32817258
- [Background] Singh SJ, Barradell AC, Greening NJ, Bolton C, Jenkins G, Preston L, Hurst JR. British Thoracic Society survey of rehabilitation to support recovery of the post-COVID-19 population. BMJ Open. 2020 Dec 2;10(12):e040213. doi: 10.1136/bmjopen-2020-040213. PMID 33268418
- [Background] Fugazzaro S, Contri A, Esseroukh O, Kaleci S, Croci S, Massari M, Facciolongo NC, Besutti G, Iori M, Salvarani C, Costi S; Reggio Emilia COVID-19 Working Group. Rehabilitation Interventions for Post-Acute COVID-19 Syndrome: A Systematic Review. Int J Environ Res Public Health. 2022 Apr 24;19(9):5185. doi: 10.3390/ijerph19095185. PMID 35564579
- [Background] Spielmanns M, Buelow MM, Pekacka-Egli AM, Cecon M, Spielmanns S, Windisch W, Hermann M. Clinical and Functional Predictors of Response to a Comprehensive Pulmonary Rehabilitation in Severe Post-COVID-19 Patients. Microorganisms. 2021 Nov 28;9(12):2452. doi: 10.3390/microorganisms9122452. PMID 34946054
- [Background] Kolodziej M, Wyszynska J, Bal-Bochenska M. COVID-19: A New Challenge for Pulmonary Rehabilitation? J Clin Med. 2021 Jul 29;10(15):3361. doi: 10.3390/jcm10153361. PMID 34362142
- [Background] Dalbosco-Salas M, Torres-Castro R, Rojas Leyton A, Morales Zapata F, Henriquez Salazar E, Espinoza Bastias G, Beltran Diaz ME, Tapia Allers K, Mornhinweg Fonseca D, Vilaro J. Effectiveness of a Primary Care Telerehabilitation Program for Post-COVID-19 Patients: A Feasibility Study. J Clin Med. 2021 Sep 27;10(19):4428. doi: 10.3390/jcm10194428. PMID 34640447
- [Background] D'Angelo E, Prandi E, Marazzini L, Milic-Emili J. Dependence of maximal flow-volume curves on time course of preceding inspiration in patients with chronic obstruction pulmonary disease. Am J Respir Crit Care Med. 1994 Dec;150(6 Pt 1):1581-6. doi: 10.1164/ajrccm.150.6.7952618.
- [Background] Koulouris N, Mulvey DA, Laroche CM, Green M, Moxham J. Comparison of two different mouthpieces for the measurement of Pimax and Pemax in normal and weak subjects. Eur Respir J. 1988 Oct;1(9):863-7. PMID 3229485
- [Background] Ringqvist T. The ventilatory capacity in healthy subjects. An analysis of causal factors with special reference to the respiratory forces. Scand J Clin Lab Invest Suppl. 1966;88:5-179. No abstract available. PMID 4283858
- [Background] Darling RC, Cournand A, Richards DW. STUDIES ON THE INTRAPULMONARY MIXTURE OF GASES. III. AN OPEN CIRCUIT METHOD FOR MEASURING RESIDUAL AIR. J Clin Invest. 1940 Jul;19(4):609-18. doi: 10.1172/JCI101163. No abstract available. PMID 16694777
- [Background] Macintyre N, Crapo RO, Viegi G, Johnson DC, van der Grinten CP, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, Gustafsson P, Hankinson J, Jensen R, McKay R, Miller MR, Navajas D, Pedersen OF, Pellegrino R, Wanger J. Standardisation of the single-breath determination of carbon monoxide uptake in the lung. Eur Respir J. 2005 Oct;26(4):720-35. doi: 10.1183/09031936.05.00034905. No abstract available. PMID 16204605
- [Background] Standardized lung function testing. Official statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:1-100. No abstract available. PMID 8499052
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- See also: Coronavirus cases — http://coronavirus.jhu.edu/map.html
- See also: Coronavirus cases — http://covid19.who.int/region/euro/country/gr

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05736939/Prot_SAP_000.pdf